CLINICAL TRIAL: NCT04809714
Title: The Role of Blood Flow Restriction Therapy in the Postop Rehabilitation of Elderly Patients With Hip Fractures: A Randomized Controlled Pilot Study
Brief Title: The Role of Blood Flow Restriction Therapy in Postoperative Elderly Patients With Hip Fracture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Clay Spitler, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300006887; UL 1 TR003096 (Other Grant/Funding Number: Foundation for Orthopaedic Trauma)
Record Dates: First submitted 2021-03-06; First posted 2021-03-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hip Fractures; Muscle Atrophy
Keywords: Hip Surgery; Geriatric; Blood flow restriction therapy; Muscle atrophy; Muscle disuse
MeSH Terms: conditions — Hip Fractures; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The control group will undergo a graduated therapy protocol that mirrors that of the intervention group except that they will use a Delfi tourniquet system blood pressure cuff with a limb occlusion pressure (LOP) of only 10%. This is compared to the intervention group that will have a therapeutic LOP of 60-100%. This means that patients will have a cuff on their limb and are thus blinded to their group allocation but the pressure is set to such a low level that no additional effect on muscle hypertrophy is expected based on prior research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Routine Post-operative Physical Therapy (Active Comparator): The control group will undergo routine post-op and undergo a modified version of the graduated therapy protocol.
  Interventions: Other: Routine Post-operative Physical Therapy
- Routine Physical Therapy + Blood Flow Restriction and Neuromuscular Electrical Stimulation (NMES) (Experimental): The intervention group will start with a Delfi tourniquet system cuff set on a limb occlusion pressure (LOP) of 60-100%. The intervention group will also use a neuromuscular electrical stimulation device at therapeutic level in addition to BFR.
  Interventions: Device: Blood Flow Restriction with Delfi Tourniquet System Cuff

INTERVENTIONS:
Device: Blood Flow Restriction with Delfi Tourniquet System Cuff — Postoperative rehabilitation will occur up to twice a day for 5 days a week for 2 weeks using a Delfi tourniquet system blood pressure cuff with a limb occlusion pressure (LOP) of 60-100%. For each physical therapy session, participants will undergo therapy following a standardized protocol of 3-5 difference exercises each with 4 sets total in addition to NMES.
  Arms: Routine Physical Therapy + Blood Flow Restriction and Neuromuscular Electrical Stimulation (NMES)
Other: Routine Post-operative Physical Therapy — The control group with undergo a post-op therapy protocol that mirrors that of the intervention group except that they will use a Delfi tourniquet system blood pressure cuff with a limb occlusion pressure (LOP) of only 10%. Participants will use a neuromuscular electrical stimulation device operating at a sub-therapeutic level.
  Arms: Routine Post-operative Physical Therapy

SUMMARY:
The investigators aim to study the use of blood flow restriction therapy (BFR) to augment routine post-operative physical therapy in elderly patients (age >= 65) after recovering from surgical treatment of hip fractures.

DETAILED DESCRIPTION:
For elderly patients, a hip fracture is a life-altering event associated with poor overall outcomes despite early surgical treatment. The elderly population and those with significant osteopenia is growing exponentially and thus the optimal treatment and rehabilitation of hip fractures warrants increased investigation. Despite numerous interventions, falls plague the elderly population and hip fractures remain a very common problem for this population that needs to be addressed. Rapid deconditioning plays a significant role in patient morbidity following hip surgery. Recently, blood flow restriction (BFR) treatment has been shown to be effective in improving muscle strength when combined with low load resistance training physical therapy programs in elderly patients. Few studies have examined BFR in post-operative orthopedic trauma patients. The investigators aim to study the use of BFR to augment post-operative physical therapy in elderly patients (age >= 65) in the first 2-weeks after recovering from surgical treatment of hip fractures. Due to the profound muscle atrophy that occurs in the immediate postoperative period because of immobility and disuse, the investigators hypothesize that BFR may provide an anabolic effect and conserve muscle strength. The investigators hypothesis was inspired by the findings of the Nobel Prize in Physiology 2019 which describes how varying levels of oxygen shape both physiology and pathology. This is a prospective, randomized blinded 2-week study of elderly patients recovering from surgical treatment of hip fractures with two arms: 1) routine post-op physical therapy 2) routine physical therapy + BFR and neuromuscular electrical stimulation (NMES) beginning on postoperative day 1 and occurring 5 days per week for 2 weeks. To optimize safety, the study will be in an inpatient-only setting and supervised by team members certified in the application of BFR. The investigators plan to apply lessons learned to a larger 8-week intervention upon completion of this short-term pilot study. To our knowledge, this is the first study to use BFR in postoperative geriatric patients. Main outcomes will include thigh leg circumference on postoperative day 1 and at the end of week 2, adverse event log for complications, knee extension strength via handheld dynamometry (HHD) at post-op day 1 and week 2, gait speed, functional tests including timed up and go, opioid MME (morphine milligram equivalent) consumption and patient perceived pain and quality of life measures. The investigators anticipate BFR therapy will be tolerated well, improve global patient health and satisfaction, lead to lower extremity muscle hypertrophy, and enhance functional recovery after geriatric hip fracture carrying tremendous potential for extramural funding and scientific advancement.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years old, any sex, any ethnicity
* Isolated, closed proximal femur fracture without any prior surgery or orthopedic implants to affected proximal femur. This includes all fractures with primary fracture line that is proximal to the lesser trochanter. For example, subtrochanteric femur fractures are excluded whereas reverse obliquity intertrochanteric femur fractures may be included.
* OTA codes 31A, 31B, and 31C
* Segmental and pathologic femur fractures are excluded.
* Ambulatory without assistive device prior to injury
* Community living prior to injury
* No injury or surgery to the contralateral lower extremity within past 1 year
* Alert and oriented and able to provide informed consent for self
* English speaking
* Able to weight bear as tolerated after surgery as deemed by treating orthopedic surgeon
* Able to tolerate light exercise (could walk approximately 0.5 mile without significant pain or shortness of breath) preoperatively as determined by patient self-reported history

Exclusion Criteria:

* Presence of other significant injuries at the time of injury to the proximal femur that would require additional surgery
* Significant delay in presentation to health care facility (>3 days from time of injury) for assessment and treatment of the proximal femur fracture
* History of DVT in any extremity, existing DVT in any extremity, or any condition known to increase risk for coagulopathy including but not exclusively current pregnancy, current diagnosis of cancer/cancer that is being treated
* Current use of any medication or supplement that may increase blood clotting risk
* History of: sickle cell anemia, peripheral arterial disease, dementia, actively treated cancer
* Varicose veins in either lower extremity
* Any significant medical condition that would preclude ability to bear weight as tolerated postoperatively
* Significant cardiac disease as defined by recent stent placement in the past year or presence of implantable pacemaker device
* Morbid obesity (BMI >40)
* Prior surgery to either lower extremity within one year
* Prior surgery or injury to either lower extremity that would preclude application of a tourniquet and includes but not exclusively: skin grafting, vascular bypass grafting, dialysis site, chronic wound, lymphotomies, varicose vein surgery, presence of tumor)
* Soft tissue injury to either lower extremity that precludes placement of tourniquet
* Diagnosis of uncontrolled hypertension (BP greater than 180/110 on at least two measurements as measured during inpatient stay before surgery)
* Patients with potentially severe problems with maintaining follow-up (ex. Patients who are prisoners, homeless at time of injury, severe dementia, intellectually challenged without adequate family support or have documented significant psychiatric disorder)
* COVID-19 positive
* Admission to ICU postoperatively
* Inadequate postop x-rays placing patient at high risk of implant-related failure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants thigh circumference measurement | At enrollment
  10cm proximal to superior pole patella and leg circumference measured at 10 distal to inferior pole patella for both extremities
Participants thigh circumference measurement | Post op 2 weeks
  10cm proximal to superior pole patella and leg circumference measured at 10 distal to inferior pole patella for both extremities
Therapist-reported compliance and adverse event logs | Post op 2 weeks
  Specify if able to perform specific exercises to completion or not
Objective muscle strength measured by a handheld dynamometer | At enrollment
  To assess strength of quadriceps extension
Objective muscle strength measured by a handheld dynamometer | Post op 2 weeks
  To assess strength of quadriceps extension
Participant self-reported outcome for pain | Post op 2 weeks
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The range of scores are from 0-100. A higher score indicates greater pain intensity.
Participant self-reported outcome: Perceived Exertion (Borg Rating of Perceived Exertion) | Post op 2 weeks
  To assess effort and exertion, breathlessness and fatigue during exercise

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | Post op 2 weeks
  Measurement of the time in seconds for a person to rise from sitting from a standard arm chair, walk 3 meters, walk back to the chair, and sit down.
Modified 30-second sit-to-stand test | Post op 2 weeks
  Measurement of the number of sit-to-stands a person can complete in 30 seconds.
Five-times sit to stand test | Post op 2 weeks
  Measures lower extremity strength and function. Participants are asked to stand up from a seated position and sit down 5 times as quickly as possible.
Functional testing performed | Post op 2 weeks
  5 Meter gait speed test
12-Item Short Form Health Survey (SF-12) (Mental Health Component) | Post op 2 weeks
  This is a general health questionnaire with higher scores representing better health. A summary score from the SF-12 (Mental Health Component) will be reported. The score may be represented as a Z-score. The average summary score is 50 points with a standard deviation of 10 points.
12-Item Short Form Health Survey (SF-12) (Physical Health Component) | Post op 2 weeks
  This is a general health questionnaire with higher scores representing better health. A summary score from the SF-12 (Physical Health Component) will be reported. The score may be represented as Z-score. The average of the summary score is 50 points with a standard deviation of 10 points.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Post op 2 weeks
  This questionnaire measures physical, mental, and social health. Higher scores represents more of the concept being measured. A score of 40 is one standard deviation lower than the mean of the reference population while a score of 60 is one standard deviation higher than the mean of the reference population.
Pain medicine requirements during 2-week stay | Post op 2 weeks
  To assess the milligram morphine equivalents of pain medicine used.

OTHER OUTCOMES:
Post-operative complications: Mortality | Post op 2 weeks
  Mortality will be assessed by living status.
Post-operative complications: Blood Clots | Post op 2 weeks
  Blood clots will be assessed by a detailed physical examination.
Post-operative complications: Deep Infection | Post op 2 weeks
  Deep infection will be assessed by the need to return to the operating room for surgical debridement or by the presence of positive cultures.
Post-operative complications: Nerve Damage | Post op 2 weeks
  Nerve damage will be assessed by a detailed physical examination assessing both sensory and motor functions.
Number of patient-reported falls | Post op 2 weeks
  To assess tolerance of BFR we will record the incidence of falls.

CONTACTS AND LOCATIONS:
Overall Officials: David A Patch, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.

REFERENCES:
- [Background] Prabhakar NR. 2019 Nobel Prize in Physiology or Medicine. Physiology (Bethesda). 2020 Mar 1;35(2):81-83. doi: 10.1152/physiol.00001.2020. No abstract available. PMID 32024429
- [Background] Bhandari M, Devereaux PJ, Swiontkowski MF, Tornetta P 3rd, Obremskey W, Koval KJ, Nork S, Sprague S, Schemitsch EH, Guyatt GH. Internal fixation compared with arthroplasty for displaced fractures of the femoral neck. A meta-analysis. J Bone Joint Surg Am. 2003 Sep;85(9):1673-81. doi: 10.2106/00004623-200309000-00004. PMID 12954824
- [Background] Simunovic N, Devereaux PJ, Sprague S, Guyatt GH, Schemitsch E, Debeer J, Bhandari M. Effect of early surgery after hip fracture on mortality and complications: systematic review and meta-analysis. CMAJ. 2010 Oct 19;182(15):1609-16. doi: 10.1503/cmaj.092220. Epub 2010 Sep 13. PMID 20837683
- [Background] Baker BS, Stannard MS, Duren DL, Cook JL, Stannard JP. Does Blood Flow Restriction Therapy in Patients Older Than Age 50 Result in Muscle Hypertrophy, Increased Strength, or Greater Physical Function? A Systematic Review. Clin Orthop Relat Res. 2020 Mar;478(3):593-606. doi: 10.1097/CORR.0000000000001090. PMID 31860546
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Proximal, Distal, and Contralateral Effects of Blood Flow Restriction Training on the Lower Extremities: A Randomized Controlled Trial. Sports Health. 2019 Mar/Apr;11(2):149-156. doi: 10.1177/1941738118821929. Epub 2019 Jan 14. PMID 30638439
- [Background] Centner C, Wiegel P, Gollhofer A, Konig D. Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. Sports Med. 2019 Jan;49(1):95-108. doi: 10.1007/s40279-018-0994-1. PMID 30306467
- [Background] Natsume T, Ozaki H, Saito AI, Abe T, Naito H. Effects of Electrostimulation with Blood Flow Restriction on Muscle Size and Strength. Med Sci Sports Exerc. 2015 Dec;47(12):2621-7. doi: 10.1249/MSS.0000000000000722. PMID 26110693